CLINICAL TRIAL: NCT02019290
Title: A SINGLE CENTER, OPEN LABEL, FIXED SEQUENCE STUDY TO INVESTIGATE THE EFFECT OF MULTIPLE DOSE BITOPERTIN ON SINGLE DOSE PHARMACOKINETICS OF MIDAZOLAM IN HEALTHY VOLUNTEERS
Brief Title: A Study Exmining the Effect of Multiple Doses of Bitopertin on the Single Dose Pharmacokinetics of Midazolam in Healthy Volunteers.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP29245
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Midazolam; (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

ARMS (1):
- bitopertin-Midazolam (Experimental)
  Interventions: Drug: Midazolam; Drug: bitopertin

INTERVENTIONS:
Drug: Midazolam — Single oral doses will be given on Days 1 and 15, after an overnight fast.
Drug: bitopertin — An oral dose will be given daily in the morning from Days 2-15. On Days 14 and 15, bitopertin will be given after an overnight fast; on Days 2-13, bitopertin will be given under fed conditions.

SUMMARY:
This will be a single-center, open-label, inpatient/outpatient, fixed-sequence study examining the effect of multiple doses of bitopertin on single doses of Midazolam in healthy volunteers.

A single oral dose on Midazolam (7.5 mg) will be administered on Day 1 after an overnight fast. Daily oral doses of bitopertin will be given under fed conditions from Days 2-13 and after fasting on Day 14. Oral doses of bitopertin and Midazolam (7.5 mg) will be co-administered on Day 15, after an overnight fast.

Pharmacokinetics will be assessed throughout. Total time on treatment is expected to be 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 to 65 years of age, inclusive.
* A BMI between 18 to 30 kg/m2, inclusive.
* Healthy as determined by the Investigator on the basis of medical/surgical history, physical examination, clinical laboratory test results, vital signs and 12-lead electrocardiogram (ECG)
* Female participants must use effective contraception as defined by the protocol and cannot be pregnant or breastfeeding
* Non-smoker or smoker of fewer than 10 cigarettes per day
* Must be able to refrain from smoking during the in-patient stay

Exclusion Criteria:

* Personal or family history of congenital long QT syndrome or family history of sudden death
* Any major illness within the 4 weeks prior to dosing or any acute disease state within 7 days prior to study start
* History of alcoholism, drug abuse or addiction within the last year prior to study start, or suspicion of drug abuse/addiction or alcohol use prior to study start
* Current alcohol consumption averaging more than 24 g of alcohol per day
* Any significant allergic reactions against any drug, or multiple allergies in the judgment of the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02-10 (Estimated); Primary Completion 2014-03-31 (Estimated); Study Completion 2014-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma area under the concentration-time curve (AUC) of midazolam after bitopertin administration | Days 1 and 15

SECONDARY OUTCOMES:
Change in 1'-hydroxymidazolam plasma AUC after bitopertin administration | Days 1 and 15
Incidence of adverse events | Approximately 76 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche